CLINICAL TRIAL: NCT04165876
Title: High Definition Transcranial Direct Current Stimulation: Effects on the Somatosensory System
Brief Title: HD-tDCS: Effects on the Somatosensory System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Danish National Research Foundation (Other)
Responsible Party: Principal Investigator, Sebastian Kold Sørensen, PhD-fellow, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: N-20180085.v1
Record Dates: First submitted 2019-09-11; First posted 2019-11-18 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Acute Pain; Neuroplasticity; Brain Modulation; Somatosensory Function
Keywords: tDCS; HD-tDCS; Somatosensory function; QST; quantitative sensory testing; Non-invasive brain stimulation; NIBS; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Longitudinal, sham-controlled, parallel groups design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The stimulation protocol is blinded and randomized using the software's "double-blinding" function.
  The subjects are randomly assigned to one of four groups receiving the corresponding stimulation protocol. One of which is a sham-stimulation (placebo), that imitates the experience of real stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Primary motor cortex (Active Comparator)
  Interventions: Device: Primary Motor Cortex Stimulation
- Dorsolateral prefrontal cortex (Active Comparator)
  Interventions: Device: Dorsolateral Prefrontal Cortex Stimulation
- Multi-modal stimulation (DLPFC+M1) (Active Comparator)
  Interventions: Device: Multimodal Stimulation (DLPFC+M1)
- Sham-stimulation (Sham Comparator)
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Primary Motor Cortex Stimulation — Using the Starstim 32, HD-tDCS equipment we provide 20 minutes of 2 mA anodal stimulation of primary motor cortex (M1) using a ring-cathode configuration
  Arms: Primary motor cortex
Device: Dorsolateral Prefrontal Cortex Stimulation — Using the Starstim 32, HD-tDCS equipment we provide 20 minutes of 2 mA anodal stimulation of dorsolateral prefrontal cortex (DLPFC) using a ring-cathode configuration
  Arms: Dorsolateral prefrontal cortex
Device: Multimodal Stimulation (DLPFC+M1) — Using the Starstim 32, HD-tDCS equipment we provide 20 minutes of 2 mA anodal multimodal stimulation of dorsolateral prefrontal cortex (DLPFC) and primary motor cortex simultaneously using ring-cathode configurations around the two anodes.
  Arms: Multi-modal stimulation (DLPFC+M1)
Device: Sham stimulation — Using the Starstim 32, HD-tDCS equipment we provide sham stimulation with 30 seconds of ramping up to 2 mA intensity, then turning off for 19 minutes and then ramping down from 2 mA intensity to 0 in the last 30 seconds.
  Arms: Sham-stimulation

SUMMARY:
The purpose of this study is to investigate the efficacy of high definition tDCS on different cortical targets in modulating the nociceptive system in the healthy subjects.

DETAILED DESCRIPTION:
The investigators aim to investigate the efficacy of different HD-tDCS electrode configurations on modulating the somatosensory/nociceptive system.

This is done to investigate the hypothesis, that different stimulation protocols can be used to modulate the somatosensory and nociceptive system, as shown in the previous studies, but that it is necessary to uncover the most efficient way to do so.

The study uses a double-blinded, sham-controlled, longitudinal design, where quantitative sensory testing will be used to assess the somatosensory function of the participants before and after a receiving a specific configuration of HD-tDCS on three consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women.
* Able to speak, read and understand English or Danish.

Exclusion Criteria:

* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Current use of opioids, antipsychotics, benzodiazepines
* Previous or current neurological, musculoskeletal, rheumatic, malignant, inflammatory or mental illnesses
* Current or prior chronic pain conditions
* Lack of ability to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Change in pressure pain threshold | Six assessments over three days: Baseline is assessed before any intervention at day one, and then the pain thresholds are assessed before and after each intervention on the subsequent two days.
  A hand-held pressure algometer (Somedic, Hörby, Sweden) with a 1-cm2 probe will be used to record the pressure pain threshold. The pressure is increased gradually at a rate of 30 kPa/s. The measurement is repeated three times on on flexor carpi radialis.

SECONDARY OUTCOMES:
Change in tactile detection threshold | Six assessments over three days: Baseline is assessed before any intervention at day one, and then the sensory thresholds are assessed before and after each intervention on the subsequent two days.
  Tactile threshold will be measured using an anaesthesiometer consisting of a set of Von Frey filaments. The filaments are made of nylon fibre of various diameters so as to provide a range of forces of up to 300 grams. The minimum force that the subject can detect will be identified. This will be assessed on flexor carpi radialis on the right hand arm.
Change in mechanical pain threshold | Six assessments over three days: Baseline is assessed before any intervention at day one, and then the sensory thresholds are assessed before and after each intervention on the subsequent two days.
  Mechanical pain threshold (MPT) will be measured using a set of weighted pinprick stimulators with a flat contact area of 0.25 mm diameter that exert forces between 8 and 512 mN. Threshold procedures will use a method of limits with up to five series of ascending and descending stimulus intensities. This will be assessed on flexor carpi radialis on the right hand arm.
Change in Thermal Sensory Detection | Six assessments over three days: Baseline is assessed before any intervention at day one, and then the sensory thresholds are assessed before and after each intervention on the subsequent two days.
  A 3×3 cm (9 cm2) contact thermode (Medoc Advanced Medical Systems, Israel) will be used to apply thermal stimulation. Each stimulus will be started at 32°C and thresholds of heat and cold sensory detection will be assessed by ascending or descending ramps in temperature to the cutoffs of 0-50 °C. This will be assessed on flexor carpi radialis on the right hand arm.
Change in Thermal Pain Detection | Six assessments over three days: Baseline is assessed before any intervention at day one, and then the sensory thresholds are assessed before and after each intervention on the subsequent two days.
  A 3×3 cm (9 cm2) contact thermode (Medoc Advanced Medical Systems, Israel) will be used to apply thermal stimulation. Each stimulus will be started at 32°C and thresholds of heat and cold pain detection will be assessed by ascending or descending ramps in temperature to the cutoffs of 0-50 °C. This will be assessed on flexor carpi radialis on the right hand arm.
Change in conditioned pain modulation (CPM) | Six assessments over three days: Baseline is assessed before any intervention at day one, and then the sensory thresholds are assessed before and after each intervention on the subsequent two days.
  A computer-controlled cuff pressure algometer (Nocitech, Denmark) with an air-filled tourniquet cuff (VBM, Germany) will be used to record cuff pressure-induced pain thresholds over the muscle bulk on the calfs. The pressure is increased gradually at a rate of 1 kPa/s to assess pain tolerance on a 0-10 VAS scale, where 0 is no pain at all and 10 is the worst pain imaginable.
  During CPM testing, the pain tolerance is first assessed on one leg marking the baseline. The pressure pain tolerance is then assessed on the same leg again, while the contralateral calf is applied a simultaneous painful pressure stimulus. The outcome of the CPM testing is the difference in pressure pain tolerance measured in kPA between the first and the second assessment. The larger the positive difference is between the baseline and the second assessment, the stronger CPM effect the subject has.
Change in vibration detection threshold. | Six assessments over three days: Baseline is assessed before any intervention at day one, and then the sensory thresholds are assessed before and after each intervention on the subsequent two days.
  Vibration detection threshold (VDT) will be determined with a Rydel-Seiffer tuning fork (64 Hz, 8/8 scale), which will be placed three times over a bony prominence of the distal part of the ulna on the right arm. Subjects are to indicate the disappearance of vibratory sensations.
Change in temporal summation of pain (TSP). | Six assessments over three days: Baseline is assessed before any intervention at day one, and then the sensory thresholds are assessed before and after each intervention on the subsequent two days.
  TSP will be applied using cuff pressure algometry. A total of 10 repeated mechanical pressure stimuli will be delivered at 0.5 Hz (1-s stimuli duration and 1-s interval between stimuli) to the test area. During the 10 repeated stimuli, subjects will continuously rate the pain intensity on a 10-cm continuous VAS. TSP is assessed on the calf of the right leg.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Graven-Nielsen, Prof., Principal Investigator — Aalborg University
Locations (1):
- Center for Neuroplasticity and Pain, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kold S, Graven-Nielsen T. Effect of anodal high-definition transcranial direct current stimulation on the pain sensitivity in a healthy population: a double-blind, sham-controlled study. Pain. 2021 Jun 1;162(6):1659-1668. doi: 10.1097/j.pain.0000000000002187. PMID 33449508